CLINICAL TRIAL: NCT03997981
Title: Chemotherapy Induced Peripheral Neuropathy Natural History Study (EPIPHANY)
Acronym: EPIPHANY
Status: Recruiting | Type: Observational
Sponsor: Disarm Therapeutics (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Eli Lilly and Company (Industry)
Other Study IDs: 18232; H7I-MC-S028 (Other: Eli Lilly and Company); 10001 (Other: Disarm Therapeutics)
Record Dates: First submitted 2019-06-12; First posted 2019-06-25 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: CIPN

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples collected for measuring biomarkers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Breast cancer patients with weekly/biweekly paclitaxel regimen
- Breast cancer patients receiving docetaxel regimen
- Lymphoma patients receiving vincristine regimen
- Multiple myeloma patients receiving bortezomib regimen
- Colorectal cancer patients receiving oxaliplatin-based regimens

SUMMARY:
This is a prospective natural history study of CIPN in approximately 200 participants receiving taxanes (paclitaxel, docetaxel) for breast cancer, bortezomib for multiple myeloma, oxaliplatin-based regimens for colorectal cancer, or vincristine for lymphoma.. Demographic data, medical history, electronic PROs, ClinROs blood biomarkers including NF-L, PGx DNA analyses and Bedside-QST will be assessed at Baseline. The Observation Period will initiate with the first dose of chemotherapy and conclude with the last dose of chemotherapy. During the Observation Period, participants will be evaluated for the development of CIPN using PROs and ClinROs. Blood biomarkers and Bedside-QST will be measured at various timepoints corresponding with treatment regimen schedules throughout the observation period. The Post Chemotherapy Follow-up Period will begin with the first visit after the last dose of chemotherapy and conclude 6 months after the last dose of chemotherapy. During the Post Chemotherapy Follow-up Period, participants will be evaluated for CIPN using PROs and ClinROs. Blood biomarkers and Bedside-QST will also be measured at the beginning and at the end of the Post-Chemotherapy Follow-up Period. PROs will be assessed electronically on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met in order to be enrolled in the study:

* Age ≥18 years
* Life expectancy ≥6 months
* Participants with Common Terminology Criteria for Adverse Events (CTCAE) Grade 0 CIPN (exception, patients with multiple myeloma treated with bortezomib, CTCAE Grade <=1)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Breast cancer only:

  * Breast cancer beginning treatment with paclitaxel or docetaxel with curative intent (i.e., not metastatic disease beyond regional lymph nodes)
  * Planned minimum of 6 cycles of chemotherapy
* Lymphoma only:

  * Incident lymphoma initiating treatment with vincristine
  * Planned minimum of 4 cycles of chemotherapy
* Oxaliplatin-based regimens, Stage III colorectal cancer: Total of 6 months (planned minimum of 12 cycles). May consider Stage IV with minimal metastatic confirmed with Sponsor prior to enrollment
* Bortezomib use in untreated multiple myeloma: Total of 4 months (planned minimum of 9 cycles)
* Written informed consent given
* Enrollment must be completed prior to receiving the first dose of chemotherapy

Exclusion Criteria:

Patients meeting ANY of the following criteria are not eligible for participation:

* Evidence of central nervous system metastases
* Evidence of clinically significant peripheral neuropathy (CTCAE >2) as defined by patient report of frequent numbness or tingling in the hands or feet
* Any uncontrolled serious illness or medical condition that would impact the conduct of the current study
* Previous exposure to neurotoxic chemotherapy drugs
* Pre-existing neurodegenerative disease (Parkinson's, Alzheimer's, Huntington's, etc.), neuromuscular disorder (multiple sclerosis, ALS, polio, hereditary neuromuscular disease) or history of stoke or history of traumatic brain injury
* General anesthesia less than one month prior to the first dose of neurotoxic chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will enroll approximately 200 participants from a total of approximately 10 sites in the United States. Each participant will participate for a duration of up to 1 year after the first dose of chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-07-03 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-09 (Estimated)

PRIMARY OUTCOMES:
Percent changes in NF-L levels from Baseline to up to 6 months after the last dose of chemotherapy | Through study completion, 2 years
  Percent changes in NF-L levels from Baseline to up to 6 months after the last dose of chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - Alpha Oncology Research LLC, DeBary, Florida
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University Medical School, St Louis, Missouri
  - Ohio State University, Columbus, Ohio
  - University of Pensylvania Hospital, Philadelphia, Pennsylvania
  - University of Vermont Medical Center, Burlington, Vermont
  - VCU Medical Center, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No